CLINICAL TRIAL: NCT05797584
Title: Valutazione Ecocardiografica Della Riserva Contrattile Del Ventricolo Destro Dopo Carico Volemico Acuto Mediante Sollevamento Passivo Delle Gambe e Durante Infusione di Dobutamina in Pazienti Affetti da Scompenso Cardiaco a Frazione d'Eiezione Ridotta (HFrEF) e Preservata (HFpEF)
Brief Title: Right Ventricular Contractile Reserve in HF
Acronym: RISE-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09C923
Record Dates: First submitted 2023-03-18; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Dobutamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EchocardiocolorDoppler (Other): EchocardiocolorDoppler examination
  Interventions: Drug: Dobutamine; Other: Passive leg raising

INTERVENTIONS:
Drug: Dobutamine — Dobutamine 5.0 - 10.0 mcg/Kg/min ev
Other: Passive leg raising — Passive leg raising for acute volume load

SUMMARY:
Right ventricle dysfunction and pulmonary hypertension are related to a worse prognosis in patients with heart failure with reduced left ventricular ejection fraction (HFrEF) or with normal left ventricular ejection fraction (HFpEF).

There is preliminary evidence however, that the responses of the right ventricle and of the pulmonary hemodynamics to stress tests (especially physical stress) may allow to prognostically stratify these patients, as these responses may bring out latent right ventricle dysfunction or a normal contractile reserve in patients with dysfunction at rest.

In view of the different pathophysiological mechanisms of the left ventricular dysfunction in HFpEF and in HFrEF, also the response and the adaptation of the righty ventricle to stress tests may be different in these two groups of patients.

In this preliminary two groups of 20 patients with HFpEF and HFrEF will be subjected to to simple stress tests: passive leg raising and inotropic stimulus with dobutamine.

This study intends to analyze, through colorDoppler echocardiography, the behaviour of the right ventricle and the pulmonary circulation during passive leg raining and infusion of dobutamine, in a cohort of patients with HFrEF or HFpEF.

The analysis will be focused on the relation between echocardiographic parameters, especially those concerning right ventricular function and pulmonary hemodynamics, thereby comparing the responses observed in HFrEF vs HFpEF.

Furthermore, correlations between the above-mentioned echocardiographic parameters and parameters of daily clinical practice will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* heart failure with reduced (EF ≤40%) or preserved (EF > 50%) ejection fraction
* echocardiographic acoustic window adequate for evaluation of outcome parameters
* presence of tricuspid insufficiency which allows assessment of pulmonary artery systolic pressure

Exclusion Criteria:

* recent myocardial infraction (<3 months) or unstable angina
* moderate o severe aortic or mitralic valve disease
* inadequate acoustic window
* significant anemia (hemoglobin <10 g/dl)
* recent heart surgery (< 3 months).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-03-20 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Right ventricle (RV) volume - Dobutamine | Baseline and at 5 minutes after Dobutamine infusion
  Change in RV volume
Ejection fraction - Dobutamine | Baseline and at 5 minutes after Dobutamine infusion
  Change in ejection fraction
Right ventricle (RV) volume - Passive leg raining | Baseline and at 1 minute after passive leg raising for acute volume load
  Change in RV volume
Ejection fraction - Passive leg raining | Baseline and at 1 minute after passive leg raising for acute volume load
  Change in ejection fraction

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Luca IRCCS Istituto Auxologico Italiano, Milan, MI, Italy